CLINICAL TRIAL: NCT06056518
Title: Prospective, Randomized Controlled Trial to Investigate the Impact of AI on Shared Decision Making in Post-kidney Transplant Care
Brief Title: Investigating the Impact of AI on Shared Decision Making in Post-kidney Transplant Care
Acronym: PRIMA-AI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Klemens Budde, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHA-PRIMA-AI
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Kidney Transplant Failure
Keywords: Kidney Transplantation; Graft Loss; Kidney Transplant Failure; Riks Prediction System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Routine Care (No Intervention): Patients in the "Routine Care" arm are will undergo regular follow-up at the kidney transplant center.
- AI-supported Care (Experimental): Patients in the "AI-supported Care" arm will undergo regular follow-up at the kidney transplant center. Treating physicians will be provided an AI-based risk prediction tool that predict 1-year risk of graft loss for patients in this group based on routine parameters.
  Interventions: Other: AI-based risk prediction for kidney graft loss

INTERVENTIONS:
Other: AI-based risk prediction for kidney graft loss — Implementation of AI-based risk prediction tool for the 1-year risk of kidney graft loss.
  Arms: AI-supported Care

SUMMARY:
This study aims to analyze the effects of AI-based risk prediction for graft loss on the frequency of conversations about the treatment after graft loss, as well as the associated shared decision making process in post-kidney transplant care in a German kidney transplant center (KTC), as perceived by the patient, their support person and the clinician/physician. Second, it aims to explore changes in patient and support person recall at 12 and 24 months follow-up. Implementation barriers and enablers will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* patients with functioning kidney allograft
* > 12 months after transplantation
* eGFR < 30 ml/min/1.73m2 according to CKD-EPI 2021 formula
* at least 18 years of age
* ability to communicate in German
* regular follow-up at kidney transplant center

Exclusion Criteria:

* multi-organ transplantation
* eGFR > 30 ml/min/1.73m2 according to CKD-EPI 2021 formula
* <= 12 months after transplantation
* less than 18 years of age
* not able to communicate in German
* no regular follow-up at kidney transplant center
* enrollment in another interventional study less than 1 month before participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All genders (male, female, and others) are eligible for this study.
Enrollment: 76 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Conversation about kidney replacement therapy after graft loss | 12 months
  Proportion of patients, with whom the necessity of kidney replacement therapy after kidney allograft loss is discussed

SECONDARY OUTCOMES:
CollaboRATE mean score after 12 months | 12 months
  CollaboRATE mean score of all study visits from study inclusion until month 12 (values 0 - 9, higher values indicating better outcome)
CollaboRATE mean score after 24 months | 24 months
  CollaboRATE mean score of all study visits from study inclusion until month 24 (values 0 - 9, higher values indicating better outcome)
Control Preferences Scale mean after 12 months | 12 months
  Mean Control Preferences Scale of all study visits from study inclusion until month 12 (values 1 - 5, higher values indicating better outcome)
Control Preferences Scale mean after 24 months | 24 months
  Mean Control Preferences Scale of all study visits from study inclusion until month 24 (values 1 - 5, higher values indicating better outcome)
Kidney replacement therapy 12 months | 12 months
  Frequency of kidney replacement therapy after graft loss 12 months
Kidney replacement therapy 24 months | 24 months
  Frequency of kidney replacement therapy after graft loss 24 months
Emergency dialysis 12 months | 12 months
  Frequency of emergency dialysis after graft loss 12 months
Emergency dialysis 24 months | 24 months
  Frequency of emergency dialysis after graft loss 24 months
Dialysis initiation via AV-shunt 12 months | 12 months
  Frequency of dialysis initiation via AV-shunt after graft loss 12 months
Dialysis initiation via AV-shunt 24 months | 24 months
  Frequency of dialysis initiation via AV-shunt after graft loss 24 months
Dialysis initiation via permanent catheter 12 months | 12 months
  Frequency of dialysis initiation via permanent catheter after graft loss 12 months
Dialysis initiation via permanent catheter 24 months | 24 months
  Frequency of dialysis initiation via permanent catheter after graft loss 24 months
Retransplantation 12 months | 12 months
  Frequency of retransplantation after graft loss 12 months
Retransplantation 24 months | 24 months
  Frequency of retransplantation after graft loss 24 months
Conversation about kidney replacement therapy after graft loss | 24 months
  Proportion of patients, with whom the necessity of kidney replacement therapy after kidney allograft loss is discussed

OTHER OUTCOMES:
Qualitative analysis of semistructured interviews | 24 months
  Qualitative analysis of semistructured interviews after 24 months
Qualitative analysis of physician-patient conversations | 24 months
  Qualitative analysis of physician-patient conversations after 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Klemens Budde, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Osmanodja B, Sassi Z, Eickmann S, Hansen CM, Roller R, Burchardt A, Samhammer D, Dabrock P, Moller S, Budde K, Herrmann A. Investigating the Impact of AI on Shared Decision-Making in Post-Kidney Transplant Care (PRIMA-AI): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Apr 1;13:e54857. doi: 10.2196/54857. PMID 38557315